CLINICAL TRIAL: NCT02296411
Title: A Multicentre, Randomised, Double-blind, Placebo-controlled, 2-way Cross-over Study to Evaluate the Efficacy and Safety of CHF 5259 (Glycopyrrolate Bromide) pMDI on Top of QVAR® pMDI for the Treatment of Patients With Uncontrolled Asthma on Low-Medium Dose of Inhaled Corticosteroids
Brief Title: Efficacy of LAMA Added to ICS in Treatment of Asthma
Acronym: ELITRA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCD-05993AB1-02; 2014-001442-16 (EudraCT Number)
Record Dates: First submitted 2014-11-14; First posted 2014-11-20 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Asthma
Keywords: Asthma, Anticholinergics
MeSH Terms: conditions — Asthma | interventions — Glycopyrrolate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CHF 5259 12.5 µg (Experimental): CHF 5259 12.5 µg: 2 inhalations bid (50µg daily dose)
  Interventions: Drug: CHF 5259 12.5 µg
- CHF 5259 placebo (Placebo Comparator): CHF 5259 placebo: 2 inhalations bid
  Interventions: Drug: CHF 5259 placebo

INTERVENTIONS:
Drug: CHF 5259 12.5 µg — comparison of CHF5259 versus placebo over 2 treatment periods of 6 weeks
  Other Names: glycopyrrolate bromide
  Arms: CHF 5259 12.5 µg
Drug: CHF 5259 placebo — comparison of CHF5259 versus placebo over 2 treatment periods of 6 weeks
  Other Names: Placebo
  Arms: CHF 5259 placebo

SUMMARY:
The purpose of this study is to evaluate the superiority of the glycopyrrolate bromide (CHF 5259 pMDI) versus placebo on top of QVAR® pMDI, in terms of lung functions parameters, as well as to assess its safety.

ELIGIBILITY:
Inclusion Criteria:

* History of asthma ≥ 5 years and diagnosed before 40 years old
* Uncontrolled asthma on low-medium doses of Inhaled CorticoSteroid (ICS) with ACQ (Asthma Control Questionnaire) ≥1.5
* Pre-bronchodilator FEV1 ≥40% and <90% of their predicted normal value
* Positive reversibility test

Exclusion Criteria:

* Pregnant or lactating women
* Diagnosis of Chronic Obstructive Pulmonary Disease (COPD)
* Patients treated for asthma exacerbation in the 4 weeks prior to study entry
* Patients who are in therapy for gastroesophageal reflux disease
* Patients who have a clinically significant cardiovascular condition

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2014-11; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
FEV1 (Forced Expiratory Volume in the first second) AUC0-12h (Area Under the Curve for 0-12 hours) normalised by time on Day 42 | Day 42

SECONDARY OUTCOMES:
Peak FEV1 (Peak of Forced Expiratory Volume in the first second ) on Day 42 | Day 42

OTHER OUTCOMES:
Adverse Events and Adverse Drug reactions | Up to 17 Weeks

CONTACTS AND LOCATIONS:
Locations (28):
- Bulgaria (7):
  - Chiesi Clinical Trial Site 0107, Rousse
  - Chiesi Clinical Trial Site 0106, Sevlievo
  - Chiesi Clinical Trial Site 0101, Sofia
  - Chiesi Clinical Trial Site 0109, Sofia
  - Chiesi Clinical Trial Site 0108, Sofia
  - Chiesi Clinical Trial Site 0102, Sofia
  - Chiesi Clinical Trial Site 0103, Sofia
- Germany (6):
  - Chiesi Clinical Trial Site 0201, Berlin
  - Chiesi Clinical Trial Site 0203, Leipzig
  - Chiesi Clinical Trial Site 0202, Leipzig
  - Chiesi Clinical Trial Site 0206, Magdeburg
  - Chiesi Clinical Trial Site 0207, Radebeul
  - Chiesi Clinical Trial Site 0208, Witten
- Italy (4):
  - Chiesi Clinical Trial Site 0306, Brescia
  - Chiesi Clinical Trial Site 0301, Pisa
  - Chiesi Clinical Trial Site 0304, Pisa
  - Chiesi Clinical Trial Site 0303, Pordenone
- Netherlands (2):
  - Chiesi Clinical Trial Site 0404, Assen
  - Chiesi Clinical Trial Site 0405, Helmond
- Poland (9):
  - Chiesi Clinical Trial Site 0501, Bialystok
  - Chiesi Clinical Trial Site 0502, Bialystok
  - Chiesi Clinical Trial Site 0503, Elblag
  - Chiesi Clinical Trial Site 0507, Krakow
  - Chiesi Clinical Trial Site 0504, Krakow
  - Chiesi Clinical Trial Site 0512, Lodz
  - Chiesi Clinical Trial Site 0510, Lodz
  - Chiesi Clinical Trial Site 0505, Wroclaw
  - Chiesi Clinical Trial Site 0506, Zgierz

IPD SHARING:
Plan to Share IPD: Yes
Chiesi commits to sharing with qualified scientific and medical Researchers, conducting legitimate research, Patient-level Data, Study-level Data, the Clinical Protocol and the full CSR, providing access to clinical trial information consistently with the principle of safeguarding commercially confidential information and patient privacy. Any shared Patient-level Data is anonymized to protect personally identifiable information.
  Chiesi access criteria and complete process for clinical data sharing is available on the Chiesi Group website.
Access Criteria: Chiesi access criteria and complete process for clinical data sharing is available on the Chiesi Group website.
URL: https://www.chiesi.com/en/chiesi-clinical-trial-data-request-portal/

REFERENCES:
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2014-001442-16